CLINICAL TRIAL: NCT04838678
Title: Sympathetic Neural Patterns and Transduction in Obesity-associated Hypertension
Brief Title: Sympathetic Transduction in Obesity-associated Hypertension (OB-HTN)
Acronym: OB-HTN
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Christopher Hearon, Assistant Instructor, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STU2020-0749
Record Dates: First submitted 2021-04-06; First posted 2021-04-09 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Hypertension; Obesity
Keywords: NPY
MeSH Terms: conditions — Hypertension; Obesity | interventions — Neuropeptide Y

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Healthy Control (Experimental): Healthy age matched controls with no history of cardiovascular disease and normal bodyweight
  Interventions: Drug: Neuropeptide Y
- Hypertensive (Experimental): Hypertensive adults who are not obese
  Interventions: Drug: Neuropeptide Y
- Obese (Experimental): Obese adults who are not hypertensive
  Interventions: Drug: Neuropeptide Y
- Obese-hypertensive (Experimental): Obese adults who are being treated for hypertension
  Interventions: Drug: Neuropeptide Y

INTERVENTIONS:
Drug: Neuropeptide Y — intra-arterial infusion of neuropeptide Y

SUMMARY:
The purpose of this study is to understand how the nervous system communicates to blood vessels to increase blood pressure during stress. The study will also investigate how hypertension and obesity influence the nervous system and vascular function. The study will involve measuring sympathetic nervous system activity and blood flow during common laboratory physiological stress protocols (e.g. hypoxia, exercise), and in response to infusion of drugs that cause vasodilation or vasoconstriction.

ELIGIBILITY:
Inclusion Criteria:

* Control - BMI<30, age 18-55
* Hypertensive - BMI<30, age 18-55, diagnosis of hypertension by 24-hour ambulatory blood pressure monitoring Obese- BMI>30, age 18-55 Obese-hypertensive- BMI>30, age 18-55, diagnosis of hypertension by 24-hour ambulatory blood pressure monitoring

Exclusion Criteria:

All groups - presence of other significant cardiovascular disease, renal disease, history of smoking, diabetes,

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-07-18 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Blood flow measured by doppler ultrasound | Acutely on the day of study
  brachial and femoral artery blood flow
Muscle sympathetic nervous system activity | Acutely on the day of study
  recording of sympathetic nervous system activity from the peroneal or radial nerve

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States